CLINICAL TRIAL: NCT01288339
Title: An Open Label, Phase II Study Assessing Potential Predictive Tumor Markers in Patients With Metastatic Colorectal Cancer and Wild Type K-RAS Tumor Treated With FOLFOX Plus Panitumumab as First-line Therapy
Brief Title: Study Assessing Potential Predictive Tumor Markers in Metastatic Colorectal Cancer
Acronym: PULSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Espanol Multidisciplinario del Cancer Digestivo (Other)
Collaborators: Amgen (Industry); TFS Trial Form Support (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEMCAD-0903; 2009-017331-18 (EudraCT Number)
Record Dates: First submitted 2010-12-24; First posted 2011-02-02 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Panitumumab + FOLFOX (DP) (Experimental): Panitumumab and FOLFOX will be administered to patients with DP (MMP7+/p-IGF-IR) once every 14 days until 6 months of treatment or until disease progression (PD) or unacceptable toxicity. If patients have not progressed after 6 months of treatment with panitumumab and FOLFOX they will continue with panitumumab monotherapy until disease progression.
  Interventions: Drug: Panitumumab + FOLFOX (DP)
- Panitumumab + FOLFOX (no-DP) (Experimental): Panitumumab and FOLFOX will be administered to patients with no-DP (MMP7+/p-IGF-IR-, MMP7-/p-IGF-IR+ or MMP7-/p-IGF-IR) once every 14 days until 6 months of treatment or until disease progression (PD) or unacceptable toxicity. If patients have not progressed after 6 months of treatment with panitumumab and FOLFOX they will continue with panitumumab monotherapy until disease progression.
  Interventions: Drug: Panitumumab + FOLFOX (no-DP)

INTERVENTIONS:
Drug: Panitumumab + FOLFOX (DP) — Panitumumab and FOLFOX will be administered to patients with DP once every 14 days until 6 months of treatment or until disease progression (PD) or unacceptable toxicity. If patients have not progressed after 6 months of treatment with panitumumab and FOLFOX they will continue with panitumumab monotherapy until disease progression.
  Arms: Panitumumab + FOLFOX (DP)
Drug: Panitumumab + FOLFOX (no-DP) — Panitumumab and FOLFOX will be administered to patients with no-DP (MMP7+/p-IGF-IR-, MMP7-/p-IGF-IR+ or MMP7-/p-IGF-IR) once every 14 days until 6 months of treatment or until disease progression (PD) or unacceptable toxicity. If patients have not progressed after 6 months of treatment with panitumumab and FOLFOX they will continue with panitumumab monotherapy until disease progression.
  Arms: Panitumumab + FOLFOX (no-DP)

SUMMARY:
To estimate the progression free survival for subjects treated with panitumumab in combination with a chemotherapy regimen of oxaliplatin, 5-Fluorouracil (5-FU) and leucovorin (FOLFOX) as first-line chemotherapy regimen for subjects with metastatic colorectal cancer with WT (wild type) KRAS according to the IGFRp (protein receptor insulin growth factor) and MMP-7 (Matrilysin) expression.

DETAILED DESCRIPTION:
By transactivation, phosphorylated insulin growth factor receptor I (p-IGF-IR) can activate epidermal growth factor receptor (EGFR). Matrilysin (MMP-7), can activate IGF-IR (insulin-like growth factor receptor ) by degrading IGFBP-3 (Insulin-like growth factor-binding protein 3) and releasing IGF-I (Insulin-like growth factor 1). Concomitant expression of MMP-7 and p-IGF-IR (using a specific monoclonal antibody (p-1316) recognizing the phosphorylated carboxy-terminal part of the IGF-IR) (DP (Double Positivity)) correlates with poor prognosis in WT KRAS patients treated with anti-EGFR antibodies plus irinotecan.The primary objective of this trial is to estimate the progression free survival (PFS) by DP (Double Positivity)immunohistochemistry (IHC) expression in patients with wild-type KRAS mCRC (metastatic colorectal cancer)treated with panitumumab and mFOLFOX6. Two groups are established by DP status (MMP7+/p-IGF-IR+ vs. MMP7+/p-IGF-IR-, MMP7-/p-IGF-IR+ or MMP7-/p-IGF-IR-). With a power of 80% and a bilateral alpha level of 0.05, assuming an accrual period of 12 months (m) and a follow-up period of 18 m, 40 patients are planned to be included in each group to detect a Hazard Ratio of 2. The median PFS of the DP group is expected to be 6 m and the total number of expected events is 56. Secondary objectives include disease control rate, duration of response, time to response and survival according the DP status. Neither interim analysis nor multiple comparison adjustment is planned.Treatment: Both groups will receive panitumumab 6 mg/kg and mFOLFOX6 every 2 weeks. If patients have not progressed after 6 m of treatment they will continue with panitumumab monotherapy until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman ≥ 18 years.
* Competent to comprehend, sign, and date an IEC-approved (Ethics Committee) informed consent form
* Histologically-confirmed metastatic adenocarcinoma of the colon or rectum by the investigator.
* Wild Type K-RAS colorectal cancer determined by the designated Central Laboratory prior to inclusion in the study in the primary tumor and/or at least one metastasis.
* At least 1 uni-dimensionally measurable lesion of at least > 10 mm with spiral CT per modified RECIST criteria 1.1. (Response Evaluation Criteria In Solid Tumors)
* Patients with the following characteristics will be included:

  1. Recurrence after adjuvant treatment with 5-fluorouracil/folinic acid or capecitabine +/- radiotherapy with a disease-free interval > than 6 months after its completion.
  2. Recurrence after adjuvant treatment with oxaliplatin +/- radiotherapy with a disease-free interval > than 12 months
  3. De novo diagnosis of the disease.
* Eastern Cooperative Oncology Group performance status of 0 or 1.
* Life expectancy ≥ 3 months
* Adequate bone marrow function
* Adequate Hepatic and metabolic functions
* Adequate Renal function
* Magnesium > LLN (Lower limit of Normal)

Exclusion Criteria:

* Patients they have received prior systemic therapy for the treatment of metastatic colorectal carcinoma.
* Prior anti-EGFr antibody therapy (eg, cetuximab) or treatment small molecule EGFr tyrosine kinase inhibitors (eg, erlotinib) or EGFR signal transduction inhibitors.
* Patients who had resection of metastatic disease
* Central nervous system/brain metastases
* Prior malignant tumor in the last 5 years, except a history of basal cell carcinoma of the skin or pre-invasive cervical cancer.
* Unresolved toxicities from prior systemic therapy that, in the opinion of the investigator, does not qualify the patient for inclusion
* Presence of peripheral neuropathy (Common Toxicity Criteria (CTC) version 3.0 > grade 1), and of serious nonhealing wound, ulcer, or bone fracture.
* Hormonal therapy, immunotherapy or experimental or approved proteins/antibodies (eg, bevacizumab) ≤ 30 days before inclusion
* Significant cardiovascular disease including unstable angina or myocardial infarction within 12 months before initiating study treatment or a history of ventricular arrhythmia.
* History of interstitial pneumonitis or pulmonary fibrosis or evidence of interstitial pneumonitis or pulmonary fibrosis on baseline chest CT scan
* Treatment for systemic infection within 14 days before initiating study treatment
* Acute or sub-acute intestinal occlusion and /or active inflammatory bowel disease or other bowel disease causing chronic diarrhea (defined as > 4 loose stools per day).
* Known positive test for human immunodeficiency virus infection, hepatitis C virus, chronic active hepatitis B infection
* Any investigational agent within 30 days before enrollment
* Subject who is pregnant or breast feeding
* Surgery (excluding diagnostic biopsy or central venous catheter placement) and/or radiotherapy within 14 days prior to inclusion in the study.
* Woman or man of childbearing potential not consenting to use adequate contraceptive precautions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2010-11-08 (Actual); Primary Completion 2015-02-13 (Actual); Study Completion 2015-02-13 (Actual)

PRIMARY OUTCOMES:
Progression-free survival time according to the MMP7 status (PFS) | 5 years
  To estimate the PFS by DP immunohistochemistry (IHC) expression in patients with wild-type KRAS mCRC treated with panitumumab and mFOLFOX6. Two groups are established by DP status (MMP7+/p-IGF-IR+ vs. MMP7+/p-IGF-IR-, MMP7-/p-IGF-IR+ or MMP7-/p-IGF-IR-).

SECONDARY OUTCOMES:
Duration of response (DOR) | 5 years
  Time from first confirmed objective response to radiologic disease progression per modified RECIST criteria.
Time to response (TTR) | 5 years
  Time from randomization date to date of first confirmed objective response
Time to treatment failure (TtTF) | 5 years
  Time from enrolment to the date the decision was made to end the treatment phase for any reason.
Objective response rate (ORR) | 5 years
  Incidence of either a confirmed CR or PR per modified RECIST criteria. CRs or PRs will be confirmed no less than 28 days after the criteria for response are first met. All subjects without a confirmed response will be considered non-responders.
Disease Control Rate (DCR) | 5 years
  Incidence of either a confirmed CR or PR or stable disease (SD) while in the treatment phase; subjects prematurely discontinuing without a post baseline tumor response assessment or subjects with an observed response that is not confirmed will be considered non-responders otherwise.
Overall Survival (OS) | 5 years
  Time from randomization date to date of death.
Time To Progression (TTP) | 5 years
  Time from randomization date to date of radiologic disease progression per modified RECIST criteria.
Duration of Stable Disease (DoSD) | 5 years
  Calculated for only those subjects with a best response of SD during the treatment period, time from enrolment to date of first observed PD or death due to PD (whichever comes first) in either the combination or monotherapy phases
Incidence and severity of AEs | 5 years
  Incidence and severity of AEs (Common Toxicity Criteria version 3.0)
Molecular predictive markers for response. | 5 years
  Molecular predictive markers for response.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Maurel, MD, Study Chair — Hospital Clinic i provincial de Barcelona; Marta Martín, MD, Principal Investigator — Hospital de la Santa Creu i Sant Pau de Barcelona; Antonia Salud, MD, Principal Investigator — Hospital Arnau de Vilanova de Lleida; Antonio Arrivi, MD, Principal Investigator — Hospital Son Llatzer de Mallorca; Xavier Hernández, MD, Principal Investigator — Intitut Català d' Oncologia (ICO) de Girona; Ólbia Serra, MD, Principal Investigator — Hospital General de l'Hospitalet de Barcelona; Carles Pericay, MD, Principal Investigator — Corporació Sanitaria Parc Taulí de Barcelona; Isabel Busquier, MD, Principal Investigator — Consorcio Hospitalario Provincial de Castellon; Carlos Fernandez-Martos, MD, Principal Investigator — Instituto Valenciano de Oncología de Valencia; Jorge Aparicio, MD, Principal Investigator — Hospital Universitario La Fe de Valencia; Maria José Safont, MD, Principal Investigator — Hospital General Universitario de Valencia; Carles Bosch, MD, Principal Investigator — Hospital Dr. Peset de Valencia; Javier Gallego, MD, Principal Investigator — Hosptial General Universitario de Elche; Alberto Carmona, MD, Principal Investigator — Hosptial Morales Meseguer; Jaume Feliu, MD, Principal Investigator — Hosptial Universitario La Paz de Madrid; Ana Ruíz, MD, Principal Investigator — Hospital de Fuenlabrada de Madrid; Enrique Casado, MD, Principal Investigator — Hospital Infanta Sofía de Madrid; Ricardo Cubedo, MD, Principal Investigator — Hospital Universitario Puerta de Hierro de Madrid; Juana Maria Cano, MD, Principal Investigator — Hosptial General de Ciudad Real; Vicente Alonso, MD, Principal Investigator — Hospital Miguel Servet de Zaragoza; Monica Jorge, MD, Principal Investigator — Hospital Xeral Cies de Vigo; Herminio Manzano, MD, Principal Investigator — Hospital Son Dureta de Mallorca; Javier Rodríguez, MD, Principal Investigator — Clínica Universitaria de Navarra; Uriel Bohn, MD, Principal Investigator — Hosptial Dr. Negrin de Las Palmas de Gran Canaria; Miriam Zorrilla, MD, Principal Investigator — Hospital de Logroño; Ruth Vera, MD, Principal Investigator — Hospital de Navarra; Carlos García, MD, Principal Investigator — Complejo Asistencial de Burgos. Hospital General Yague; Santiago Albiol, MD, Principal Investigator — Hospital de l'Esperit Sant de Barcelona; José Carlos Méndez, MD, Principal Investigator — Centro Oncológico de Galicia (La Coruña); Francisco Javier Ramos, MD, Principal Investigator — Hospital de Sant Pau i Santa Tecla de Tarragona
Locations (30):
- Spain (30):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Son Espases de Mallorca, Palma de Mallorca, Balearic Islands
  - Hosptial Son Llatzer de Mallorca, Palma de Mallorca, Balearic Islands
  - Hosptial General de l'Hospitalet de Barcelona, L'Hospitalet de Llobregat, Barcelona
  - Corporació Sanitaria Parc Taulí de Barcelona, Sabadell, Barcelona
  - Hospital de l'Esperit Sant, Santa Coloma de Gramenet, Barcelona
  - Consorcio Hospitalario Provincial de Castellon, Castellon, Castellon
  - Hosptial de Logroño, Logroño, La Rioja
  - Hospital Universitario La Paz de Madrid, Madrid, Madrdi
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Hospital de Navarra, Pamplona, Navarre
  - Hospital Xeral Cies de Vigo, Vigo, Pontevedra
  - Centro Oncológico de Galícia, A Coruña
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau de Barcelona, Barcelona
  - Complejo Asitencia de Burgos. Hospital General Yague, Burgos
  - Hospital General de Ciudad Real, Ciudad Real
  - Institut Català d'Oncologia (ICO) de Girona, Girona
  - Hosptial Dr. Negrin de Las Palmas de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital Arnau de Vilanova de Lleida, Lleida
  - Hospital Infanta Sofía de Madrid, Madrid
  - Hospital Universitario Puerta de Hierro de Madrid, Madrid
  - Hospital de Fuenlabrada de Madrid, Madrid
  - Hospital Morales Meseguer, Murcia
  - Hosptial de Sant Pau i Santa Tecla de Tarragona, Tarragona
  - Hospital La Fe de Valencia, Valencia
  - Instituto Valenciano de Oncología de Valencia, Valencia
  - Hospital General de Valencia, Valencia
  - Hospital Dr. Peset de Valencia, Valencia
  - Hospital Miguel Servet de Zaragoza, Zaragoza

REFERENCES:
- [Derived] Maurel J, Alonso V, Escudero P, Fernandez-Martos C, Salud A, Mendez M, Gallego J, Rodriguez JR, Martin-Richard M, Fernandez-Plana J, Manzano H, Mendez JC, Zanui M, Falco E, Gil-Raga M, Aparicio J, Feliu J, Garcia-Albeniz X, Torres F, Rojo F, Bellosillo B, Mendiola M, Fernandez V, Reig O, Claes B, Maertens G, Sablon E, Jacobs B, Montagut C. Clinical Impact of Circulating Tumor RAS and BRAF Mutation Dynamics in Patients With Metastatic Colorectal Cancer Treated With First-Line Chemotherapy Plus Anti-Epidermal Growth Factor Receptor Therapy. JCO Precis Oncol. 2019 Dec;3:1-16. doi: 10.1200/PO.18.00289. PMID 35100697